CLINICAL TRIAL: NCT00877955
Title: Open-label, Randomized, Single-dose, 2-way Crossover Bioequivalence Study Comparing A New Alprazolam Sublingual Tablet Formulation To A Reference Alprazolam Sublingual Tablet
Brief Title: Bioequivalence Of A Test Alprazolam Sublingual Formulation Compared To A Commercial Sublingual Formulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131019
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: bioequivalence; pharmacokinetic; alprazolam; sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- alprazolam sublingual tablet reference (Active Comparator)
  Interventions: Drug: alprazolam sublingual tablet commercial
- alprazolam sublingual tablet test (Experimental)
  Interventions: Drug: alprazolam sublingual tablet test

INTERVENTIONS:
Drug: alprazolam sublingual tablet commercial — 0.5 mg sublingual tablet, single dose
  Arms: alprazolam sublingual tablet reference
Drug: alprazolam sublingual tablet test — 0.5 mg tablet, single dose
  Arms: alprazolam sublingual tablet test

SUMMARY:
This study tests the assumption that the bioavailability of alprazolam from a new sublingual formulation is the same as that from sublingual formulation expected to be used commercially in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* BMI 17.5 - 30.5
* Must provide informed consent

Exclusion Criteria:

* Clinically significant disease
* Narrow angle glaucoma
* Positive drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Alprazolam bioavailability assessed as area under the concentration-time curve (AUC) and maximum concentration (Cmax) | 11 days

SECONDARY OUTCOMES:
Alprazolam time of maximum concentration (Tmax) and half life | 11 days
Adverse events, clinical laboratory tests, vital signs | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131019&StudyName=Bioequivalence%20Of%20A%20Test%20Alprazolam%20Sublingual%20Formulation%20Compared%20To%20A%20Commercial%20Sublingual%20Formulation